CLINICAL TRIAL: NCT05316324
Title: A Randomized Controlled Trial of Prepectoral Breast Reconstruction With and Without Acellular Dermal Matrix
Brief Title: A Study of the Use of Acellular Dermal Matrix for Breast Reconstruction
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The Plastic Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-071
Record Dates: First submitted 2022-03-23; First posted 2022-04-07 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Acellular Dermal Matrix; Breast Reconstruction; Mastectomy; 22-071
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prepectoral Breast Reconstruction with ADM (Experimental)
  Interventions: Procedure: Prepectoral Breast Reconstruction with Acellular Dermal Matrix (ADM)
- Prepectoral Breast Reconstruction without ADM (Experimental)
  Interventions: Procedure: Prepectoral Breast Reconstruction without Acellular Dermal Matrix (ADM)

INTERVENTIONS:
Procedure: Prepectoral Breast Reconstruction with Acellular Dermal Matrix (ADM) — Prepectoral Breast Reconstruction with (ADM)
  Arms: Prepectoral Breast Reconstruction with ADM
Procedure: Prepectoral Breast Reconstruction without Acellular Dermal Matrix (ADM) — Prepectoral Breast Reconstruction without ADM
  Arms: Prepectoral Breast Reconstruction without ADM

SUMMARY:
The researchers are doing this study to look at the number of complications that occur immediately after prepectoral breast reconstruction when Acellular Dermal Matrix (ADM) is used compared to when ADM is not used. These complications include infections, the need for Tissue Expander (TE) or implant removal, and other conditions that lead to additional surgery.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 21-60 years
* Planning to undergo unilateral or bilateral mastectomy, prophylactically or to treat breast cancer
* Planning to undergo immediate two-stage prosthetic breast reconstruction with TE placement as the first stage
* Planning to undergo nipple-sparing or skin-sparing mastectomy
* Adequate mastectomy skin perfusion or adequate perfusion but nonviable mastectomy skin that can be excised (≤4 cm) at the defect margins with otherwise adequate perfusion
* Intraoperative confirmation of prepectoral plane viability by operating physician

Exclusion Criteria:

* History of radiotherapy to the operative breast
* Current smoker
* Non-English speaking patients
* Planning to undergo direct-to-implant reconstruction
* Prior sternotomy

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 353 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who experience major complications | 90 days
  Listed below are definitions for 90-day major complications for TEs (i.e., infection, explantation, and reoperation for any cause, including mastectomy flap necrosis):
  * Infection defined as:
  * Any event requiring the restart of antibiotics (oral or intravenous) after completion of initial perioperative antibiotics
  * Admission to the hospital for signs and symptoms of cellulitis (redness on breast mound) requiring antibiotics
  * Purulent drainage from the surgical site or incision
  * Explantation defined as the need for removal of a TE for any cause
  * Reoperation defined as skin excision performed in either the clinic or the operating room for mastectomy skin flap necrosis, surgical incision dehiscence, pending skin breakdown or another surgical complication

SECONDARY OUTCOMES:
Estimate rates of minor complications (specifically seroma) | 90 days
  Minor complication for (Tissue Expanders) TEs are defined as:
  o Seroma: Clinically significant noninfected fluid collection requiring either needle aspiration or drain replacement

CONTACTS AND LOCATIONS:
Overall Officials: Evan Matros, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm